CLINICAL TRIAL: NCT05697029
Title: Tetrandrine Tablets Used in Hospitalized Adults With COVID-19: a Double-blind, Placebo-controlled, Randomised Trial
Brief Title: Tetrandrine Tablets Used in Hospitalized Adults With COVID-19
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the lack of funding from the sponsor, the research drug and placebo cannot be obtained.
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Sun Yongchang, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2023002
Record Dates: First submitted 2023-01-21; First posted 2023-01-25 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tetrandrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tetrandrine group (Experimental): Tetrandrine 60mg TID for 28 days
  Interventions: Drug: Tetrandrine
- placebo group (Placebo Comparator): placebo TID for 28 days
  Interventions: Drug: Tetrandrine

INTERVENTIONS:
Drug: Tetrandrine — tetrandrine TID for 28 days

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of tetrandrine tablets in preventing the progression of COVID-19 from severe to critical.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effectiveness of tetrandrine tablets in preventing the progression of COVID-19 from severe to critical. The secondary objective is to evaluate the clinical indicators of COVID-19 with tetrandrine tablets treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent form voluntarily for the trial.
2. Male or female aged between 18 and 85 years (inclusive).
3. Clinically or laboratory confirmed COVID-19 within the past 7 days, as determined by a positive RT-PCR test or a positive antigen test.
4. Under resting conditions, oxygen saturation ≤93% when breathing air, or P/F value ≤ 300 mmHg (1 mmHg = 0.133 kPa).
5. No birth plan and must agree to take effective contraceptive methods.

Exclusion Criteria:

1. Received a vaccine within 4 weeks prior to the study, or plan to receive a vaccine during the study period, or received treatment with tetrandrine tables prior to enrolling in the study.
2. Patient must be on invasive mechanical ventilation/ECMO at baseline.
3. Any clinically important serious diseases unstable or uncontrolled.
4. Allergy history to any biological or other agent.
5. Patient has severe mental or psychological abnormalities, cognitive impairment or intellectual disability before being diagnosed with COVID-19.
6. Subjects who are pregnant or breastfeeding, or plan to become pregnant during the study.
7. Investigator think the subject should not participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosed with critical COVID-19 pneumonia | 84 days
  Diagnosed with COVID-19 pneumonia according to the criteria and meeting one of the following conditions: a. respiratory failure requiring mechanical ventilation, b. shock, c. other organ dysfunction requiring ICU management.

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Sun, M.D., Principal Investigator — Peking University 3rd Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No